CLINICAL TRIAL: NCT03152474
Title: Adrenal Cortical Function and Vitamin A Deficiency in Sepsis, Severe Sepsis and Septic Shock: Prospective Randomized, Double Blind Placebo Controlled Clinical Trials
Brief Title: Adrenal Cortical Function and Vitamin A Deficiency in Sepsis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7476-01; 7680-01 (Other: Los Angeles Biomedical Research Institute); 7681-01 (Other: Los Angeles Biomedical Research Institute); 7682-01 (Other: Los Angeles Biomedical Research Institute)
Record Dates: First submitted 2017-04-07; First posted 2017-05-15 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Methylprednisolone Hemisuccinate; Vitamin A

STUDY DESIGN:
Intervention Model Description: Double Blind Placebo Controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind (to investigator, subject, hospital care team and study team members except for research pharmacist), Randomized, Placebo Controlled Clinical Trial; Placebos were wrapped in foil and coded to prevent identification of study material.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Solumedrol 20mg (Active Comparator): Solumedrol injection will be given in the vein every 8 hrs. for 7 days.
  Interventions: Drug: Solumedrol 20mg; Other: Placebo
- Vitamin A 100,000 IU (Active Comparator): Vitamin A injection will be given in the arm muscle for 7 days.
  Interventions: Drug: Vitamin A 100,000 IU; Other: Placebo
- Placebo (Placebo Comparator): Placebo will be given in the vein every 8 hrs. for 7 days or given in the arm muscle for 7 days.
  Interventions: Drug: Solumedrol 20mg; Drug: Vitamin A 100,000 IU

INTERVENTIONS:
Drug: Solumedrol 20mg — Dosed Intravenous every 8 hrs.
  Other Names: Methylprednisolone Sodium Succinate
  Arms: Placebo; Solumedrol 20mg
Drug: Vitamin A 100,000 IU — Dosed Intramuscular once daily
  Other Names: Retinol
  Arms: Placebo; Vitamin A 100,000 IU
Other: Placebo — Placebo dosed intravenous every 8 hrs. or Intramuscular once daily.
  Arms: Solumedrol 20mg; Vitamin A 100,000 IU

SUMMARY:
The study involves the participant to receive a 250 mcg Cortrosyn (ACTH) Stimulation Test to test the ability of the body to make Cortisol. If the body is not able to make large amount of Cortisol (Delta Cortisol < 13 mg/dl) from the stimulation test, then the participant will be given additional cortisol like medicine called Solumedrol or matching placebo.

If the body is able to make large amounts of Cortisol (> 13 mg/dl), then the participant will receive daily shots of Vitamin A for 7 days or matching placebo.

If the participant does not respond to the stimulation test, and meets the criteria for Cortisol deficiency (all 3 cortisol concentrations < 20 mg/dl), then he/she will screen failed for the study and will be offered hydrocortisone as part of routine care by the treating physician.

DETAILED DESCRIPTION:
The eligible patients will have Sepsis, Severe Sepsis or Septic Shock. The potential subject will be approached for the study participation and if agreed will sign an Inform Consent. Patients unable to give consent, a waiver of consent was used. The participant to receive a Cortrosyn Stimulation Test to test the ability of the body to make Cortisol. The Cortrosyn Stimulation Test involves an injection into the vein in the arm. Two tablespoons of blood is collected just before the injection of Cortrosyn (250 mcg of ACTH) and again 30 minutes and 60 minutes after the injection. The results of test are available about 3 hours after the start of the test. Depending on the results of the test, subject will be either screen failed or will either receive Solumedrol or Vitamin A. Also at the beginning of the study, the amount of water in the subject's body will be measured using a machine called Impedance Monitor.

If the body is not able to make large amount of Cortisol from the stimulation test (delta increase in cortisol < 13 mg/dl), then the participant will be given additional cortisol like medicine called Solumedrol (20 mg) by injection into a vein every 8 hours for 7 days or matching placebo.

If the body is able to make large amounts of Cortisol (delta cortisol response > 13 mg/dL), then the participant will receive daily shots of Vitamin A or matching placebo for 7 days by injection into arm muscle. After 1, 3, 8 and 14 days of the study, a blood draw will performed to measure the amount of Vitamin A in the blood. Also, the urine will be collected to measure Vitamin A levels on day 1, 2, 3, 8 and 14. The ACTH stimulation test was repeated on Day 8.

The total amount of blood drawn for the study will be about 18 tablespoons.

If the participant does not respond to the stimulation test, and meets the criteria for Cortisol deficiency (All cortisol concentrations < 20 mg/dl) , then he/she will screen failed for the study and will be offered 100 mg of hydrocortisone treatment (100 mg IV every 8 hours) as part of routine care by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis
* Severe Sepsis
* Septic Shock

Exclusion Criteria:

* On glucocorticoids
* On Vitamin A
* On any active medical research study
* Failed ACTH stimulation test (All serum cortisol concentrations < 20 mg/dl)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 1993-02; Primary Completion 2000-01 (Actual); Study Completion 2000-01 (Actual)

PRIMARY OUTCOMES:
28 days mortality | 28 days
  Document the 28 days of mortality

SECONDARY OUTCOMES:
14 day mortality | 14 days
  Mortality at day 14
Number of Secondary Infections | Day 28
  Document the number of secondary infections
Days in ICU | Day 14 and Day 28
  Document the days in ICU
Number of days on ventilator | 28 days
  Document the days on ventilator
Number of days of ventilator adjusted for mortality | 28 days
  Document the number of days of ventilator adjusted for mortality
Number of days on pressor agents | 28 days
  Document the number of days on pressor agents
Number of Days on PPI or H2 blockers | 28 days
  Document the days on PPI or H2 blockers
Number of days of pressor agents corrected for mortality | 28 days
  Document the number of days of pressor agents corrected for mortality
Change in serum albumin concentration | 28 days
  Document the serum albumin concentration
New Onset Renal Failure | Day 14
  Document any new onset renal failure
Serum vitamin A concentration | baseline and day 14
  Document levels of serum vitamin A concentration
Urine Vitamin A Concentration | baseline and day 14
  Document levels of vitamin A concentration in urine
APACHE Score | Day 1 and Day 14
  Calculate and document APACHE score
ACTH Stimulation Test | Day 1 and Day 8
  Efficiency of ACTH stimulation test

IPD SHARING:
Plan to Share IPD: Yes
Only the de-identified study data will be shared with the other researchers.

REFERENCES:
- [Derived] Cherukuri L, Gewirtz G, Osea K, Tayek JA. Vitamin A treatment for severe sepsis in humans; a prospective randomized double blind placebo-controlled clinical trial. Clin Nutr ESPEN. 2019 Feb;29:49-51. doi: 10.1016/j.clnesp.2018.10.011. Epub 2018 Nov 17. PMID 30661700